CLINICAL TRIAL: NCT01800071
Title: A Cancer Research UK (CR-UK) Phase Ib Trial to Determine the Safety, Tolerability and Immunogenicity of Extended Schedule Vaccination With MVA-EBNA1/LMP2 in Patients With Epstein Barr Virus Positive (EBV+) Nasopharyngeal Carcinoma (NPC).
Brief Title: A Phase Ib Trial of MVA-EBNA1/LMP2 Vaccine in Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cancer Research UK (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CRUKD/13/001
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Nasopharyngeal Cancer; Epstein Barr Virus Infections
Keywords: Nasopharyngeal cancer; Epstein Barr Virus Infections; Vaccination
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Epstein-Barr Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MVA-EBNA1/LMP2 vaccine

SUMMARY:
This clinical study is looking at a vaccine called MVA-EBNA1/LMP2. This is a new vaccine that has already been studied in small number of cancer patients.

The vaccine is designed to boost a patient's immunity against a common virus. The virus is called Epstein Barr virus or EBV. EBV is sometimes found inside cancer cells and is commonly found in nasopharyngeal cancer cells.

DETAILED DESCRIPTION:
The main aims of the clinical study are to find out more about how the immune system responds to the vaccine, more about the potential side effects of the vaccine and the effects of giving an additional booster vaccination on the immune system.

Approximately 18 patients with EBV positive nasopharyngeal cancer (NPC) will be recruited to the trial. Patients will receive up to four vaccinations with the MVA-EBNA1/LMP2 vaccine. The first three vaccines will be given at 3 weekly intervals, followed by a fourth vaccine 12 weeks later. The vaccine will be given by intradermal injection with the dose divided across multiple injection sites on the arm, or on the thigh.

Patients will participate in the study for approximately 12 months from first vaccination and attend hospital approximately 11 times during this period. Standard safety assessments will be performed throughout the trial and at each clinic visit patients will be asked to provide research blood samples. These samples will be used to monitor the effects of the vaccine on the patient's immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed NPC in which the presence of EBV has been confirmed in the tumour by immunohistochemistry for viral antigens or EBV early RNA (EBER) fluorescent in situ hybridisation (FISH).
2. Patients in remission or with current disease for whom no standard therapy is currently appropriate or required.
3. Patients who have received primary treatment for their malignancy (radiotherapy ± chemotherapy) and up to one additional second-line course of therapy.
4. Life expectancy of at least 6 months.
5. World Health Organisation (WHO) performance status of 0 or 1 (Appendix 1).
6. Haematological and biochemical indices within the ranges shown below. These measurements must be performed within one week (Day -7 to Day 1) before the patient receives their first vaccination with MVA-EBNA1/LMP2.

   Laboratory Test Value required Haemoglobin (Hb) ≥10.0 g/dL, Lymphocyte count ≥0.5 x 10^9/L after ≥ 6 weeks have elapsed from completion of chemotherapy, Absolute neutrophil count (ANC) ≥1.0 x 10^9/L, Platelet count ≥ 75 x 10^9/L, Serum bilirubin ≤1.5 x upper limit of normal (ULN), Alkaline phosphatase (ALP) AND alanine aminotransferase (ALT) OR aspartate aminotransferase (AST) ≤ 2.5 x ULN, Calculated creatinine clearance ≥50 mL/min (uncorrected value)
7. 18 years or over.
8. Written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.

Exclusion criteria

1. Radiotherapy, chemotherapy, endocrine therapy, immunotherapy or investigational medicinal products within 6 weeks prior to trial entry.
2. Patients who, in the opinion of the investigator and multidisciplinary team managing the patient, may require another oncological treatment within 14 weeks of the first vaccination.
3. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or Grade 1 toxicities, which in the opinion of the Investigator and the Sponsor should not exclude the patient.
4. Current active auto-immune disease requiring therapy.
5. Current active eczema requiring therapy.
6. Allergy to eggs or egg products.
7. History of anaphylaxis or severe allergy to previous vaccinations or medications. Patients with a documented history of allergy to gentamicin should be discussed with the Sponsor prior to trial entry.
8. Previous splenectomy or splenic radiation, or with known splenic dysfunction.
9. Receiving current immunosuppressive medication including systemic use of corticosteroids. Prophylactic use of inhaled steroids is permitted.
10. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrolment and agree to use two highly effective forms of contraception (oral, injected or implanted hormonal contraception and condom, have a intra-uterine device and condom, diaphragm with spermicidal gel and condom) during the trial and for six months afterwards are considered eligible.
11. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of highly effective contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
12. Major thoracic or abdominal surgery from which the patient has not yet recovered.
13. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
14. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
15. History of Unstable Angina Pectoris or Myocardial Infarction up to 6 Months prior to trial entry.
16. Any other condition which in the Investigator"s opinion would not make the patient a good candidate for the clinical trial.
17. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase Ib study of MVA-EBNA1/LMP2. Participation in an observational trial would be acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Immune response to three cycles of MVA-EBNA1/LMP2 vaccine | pre-vaccination to 4 weeks post third vaccine
  To be determined by ex vivo ELIspot assays quantifying EBV EBNA1 and LMP2-specific effectors in samples before vaccination, during the three cycle vaccine course and within 4 weeks after the third vaccine cycle.
Occurrence of adverse events defined according to NCI CTCAE version 4.02 | 12 months

SECONDARY OUTCOMES:
Immune memory and recall response to MVA-EBNA1/LMP2 vaccination | pre and post vaccines one and four.
  To be determined by ex vivo ELIspot assays quantifying EBV EBNA1 and LMP2-specific effectors in samples before and within 4 weeks after the first and fourth vaccine cycles
Measurement of EBV genome levels in plasma before, during and after vaccination | pre- vaccination to 12 months post vaccination
Tumour response as determined by Immune-Related Response Criteria (irRC) | 6 months

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - University of Birmingham, Edgbaston, Birmingham
  - Royal Marsden Hospital, Fulham Road, London
  - Velindre Cancer Centre, Cardiff
  - The Beatson West of Scotland Cancer, Glasgow
  - The Christie Hospital, Manchester